CLINICAL TRIAL: NCT04706117
Title: Self-retaining Bicanalicular Intubation Stent Versus Bicanalicular Silicone Tube for Management of Canalicular Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Zamzam Mohamed alham khalil, Doctor at opthalmology department, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bicanalicular intubation
Record Dates: First submitted 2021-01-05; First posted 2021-01-12 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-12

CONDITIONS: Canalicular Obstruction
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Canalicular obstruction (Other)
  Interventions: Device: Self-retaining bicanalicular intubation stent

INTERVENTIONS:
Device: Self-retaining bicanalicular intubation stent — self-retaining bicanaliculs intubation setII(SRSII) which is the latest innovation in the field as these silicone stent segments traverse both canaliculi till the lacrimal sac. In which each end of this semicircular device has 2 stout angulated wings/flanges which pose no resistance while proceeding forward into the canaliculus, but once they get into open cavity (lacrimal sac), the flanges open up and give resistance to their removal against the common canalicular opening

SUMMARY:
The aim of the study is to evaluate outcomes of the use of self_retaining intubation set versus bicanalicular silicone tube in management of canalicular obstruction

DETAILED DESCRIPTION:
Epiphora is a condition due to obstruction of lacrimal passages either proximal or distal. Canalicular obstruction is a condition in which the lacrimal canaliculi are narrowed or occluded. Canalicular obstructions can be anatomically classified as proximal type in which the obstruction found at the initial 2-3 mm from the punctal opening while in mid canalicular type obstruction at 3-8 mm from the punctum and the distal type in which a membrane of the common canaliculs to the lacrimal sac. Canalicular obstruction can be acquired or congenital. Acquired canalicular obstruction may result from infectious and inflammatory eyelid disorders, ocular surface disease, systemic or topical medications, irradation, iatrogenic, intrinsic cannalicular tumors and trauma. The correct chioce of the techinque for given canalicular obstruction and therefore the long-term success depends on the site and degree of the obstruction, incomplete obstruction or stenosis can be treated with canalicular stenting. Proximal and mid canalicular obstructions need reconstruction by excising the focal canaliculus obstruction near the punctum and the cut ends of the canaliculus can be anastomosed over a stent. Dacryocystorhinostomy with retrograde intubation of the lacrimal system has shown some success may avoid the need for a Jones tube. Patients with symptomatic distal canalicular obstruction should undergo timely insertion of a bicanalicular silicon stent to prevent permanent and complete closure of the canaliculi. There are several modalities of canalicular intubation for the patients with distal canalicular obstruction. In patients with nasolacrimal duct and canalicular obstruction ,preferred procedures include dacryocystorhinstomy with bicanalicular or monocanalicular intubation .However,in patients with canalicular obstruction without nasolacrimal duct obstruction use bicanalicuar silicone intubation. In 2014 P.Bige' designed self-retaining bicanaliculs intubation setII(SRSII) which is the latest innovation in the field as these silicone stent segments traverse both canaliculi till the lacrimal sac. In which each end of this semicircular device has 2 stout angulated wings/flanges which pose no resistance while proceeding forward into the canaliculus, but once they get into open cavity (lacrimal sac), the flanges open up and give resistance to their removal against the common canalicular opening.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epiphora due to distal canalicular obstruction.

Exclusion Criteria: patients with epiphora due to

* Punctual stenosis
* lid malposition
* Intra-operative nasolacrimal duct obstruction
* previous eyelid or lacrimal drainage surgery
* untreated conjunctivitis, blepharitis. Dacrocystitis Proximal and mid canalicular obstruction.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of SRSll and bicanalicular silicone tube in management of canalicular obstruction | Baseline
  compare improvement of epiphora according to Munk scale for epiphora grading Grade 0 No epiphora Grade 1 Epiphora requiring dabbing less than twice a day Grade 2 Epiphora requiring dabbing 2-4 times a day Grade 3 Epiphora requiring dabbing 5-10 times a day Grade 4 Epiphora requiring dabbing more than 10 times a day Grade 5 Constant epiphora And fluorescein dye disappearance test was graded according to Ozgur et al., scale according the time of dye clearance Grade 1 <3 minutes Grade 2 3-5 minutes Grade 3 >5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Elshafei, Study Director — Minia University; Raafat M Abdelrahman, Study Director — Minia University; Amr A Mohrmed, I, Study Director — Minia University